CLINICAL TRIAL: NCT01086891
Title: Efficacy of Two Liquid Oxygen Devices in Deambulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 07/060/793
Record Dates: First submitted 2010-02-03; First posted 2010-03-15 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2012-05

CONDITIONS: To Determine the Efficacy of Two Liquid Oxygen Device

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Patients with chronic obstructive pulmonary disease who show arterial oxygen desaturation to effort.
  Interventions: Device: Oxygen conserving devices
- 2 (Experimental): Patients with interstitial lung disease who show arterial oxygen desaturation to effort
  Interventions: Device: Oxygen conserving devices

INTERVENTIONS:
Device: Oxygen conserving devices — Three 6MWT test will be performed at random with conventional oxygen continuous-flow,by Oxymizer Pendant and demand valve system. The percentage of patients correcting their desaturation and patients' acceptance of every method will be determinated.
  Other Names: Oxygen conserving devices in COPD.
  Arms: 1
Device: Oxygen conserving devices — Three 6MWT test will be performed at random with conventional oxygen continuous-flow,by Oxymizer Pendant and demand valve system. The percentage of patients correcting their desaturation and patients' acceptance of every method will be determinated
  Other Names: Oxygen conserving devices in interstitial lung disease.
  Arms: 2

SUMMARY:
Some oxygen conserving devices have been developed to diminish oxygen expense. These devices offer optimisation of oxygen therapy for deambulation by improving time autonomy of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with arterial oxygen desaturation to effort.
* COPD with TLC > 90%
* EPID with TLC < 90% and FEV1/FVC > 70%

Exclusion Criteria:

* Patients with long-term oxygen therapy (LTOT) in deambulation.
* Not clinically stable during last month.
* Smokers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-04; Primary Completion 2010-01 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
To determine the efficacy of correcting desaturation during effort and the acceptance of two different oxygen conserving devices during deambulation,one system with reservoir an another one with oxygen demand valve. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Sergi Marti, Doctor, Principal Investigator — H.Vall d'Hebron
Locations (1):
- Fundacio Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Marti S, Pajares V, Morante F, Ramon MA, Lara J, Ferrer J, Guell MR. Are oxygen-conserving devices effective for correcting exercise hypoxemia? Respir Care. 2013 Oct;58(10):1606-13. doi: 10.4187/respcare.02260. Epub 2013 Mar 19. PMID 23513249